CLINICAL TRIAL: NCT00809146
Title: A Double-blind Randomized Clinical Trial of the Efficacy of IM Midazolam Versus IV Lorazepam in the Pre-hospital Treatment of Status Epilepticus by Paramedics
Brief Title: Paramedic Treatment of Prolonged Seizures by Intramuscular Versus Intravenous Anticonvulsant Medications
Acronym: RAMPART
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Robert Silbergleit (Other)
Collaborators: Medical University of South Carolina (Other); University of California, San Francisco (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Robert Silbergleit, Principal Investigator, Professor, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01NS053031; 5U01NS056975-02 (NIH)
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Results first posted 2012-04-13 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-05

CONDITIONS: Status Epilepticus
Keywords: Status Epilepticus; Emergency Medical Services; Anticonvulsants; Drug Administration Routes; Seizures
MeSH Terms: conditions — Status Epilepticus; Seizures | interventions — Lorazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intramuscular (IM) anticonvulsant (Active Comparator): This group gets active treatment with an anticonvulsant by the intramuscular route of administration.
  Interventions: Drug: Intramuscular route of active treatment
- Intravenous (IV) anticonvulsant (Active Comparator): This group gets active treatment with an anticonvulsant by the intravenous route of administration.
  Interventions: Drug: Intravenous route of active treatment

INTERVENTIONS:
Drug: Intramuscular route of active treatment — IM administration by autoinjector of midazolam 5 mg for subjects under estimated weight of 40 kg or midazolam 10 mg for subjects with estimated weight of 40 kg or above, IV administration of matching volume of IV flush.
  Other Names: Autoinjector
  Arms: Intramuscular (IM) anticonvulsant
Drug: Intravenous route of active treatment — IV administration of lorazepam 2 mg for subjects under estimated weight of 40 kg or midazolam 4 mg for subjects with estimated weight of 40 kg or above, IM administration by autoinjector of matching volume of saline.
  Other Names: Ativan
  Arms: Intravenous (IV) anticonvulsant

SUMMARY:
The goal of this non-inferiority trial is to determine which type of routine care is the best for paramedics to stop someone from seizing.

DETAILED DESCRIPTION:
Seizures are a common medical problem. Although they can be frightening to watch, most seizures are brief and stop by themselves. Seizures that don't stop in seconds or minutes are a dangerous life-threatening medical emergency. Paramedics often have medications that can stop seizures, but the best way to give the medicines is not known. Paramedics often give medicine directly into a vein, which is called intravenous (IV) administration. This works well, but can be hard to do in a person who is seizing. It can also take some time and delay treatment. Another way to give the medicine is as a shot given into a muscle, which is called intramuscular (IM) administration. Giving the medicine this way is faster, but it may not stop the seizure as quickly.

This clinical trial, the Rapid Anti-convulsant Medication Prior to ARrival Trial (RAMPART), is designed to figure out whether giving anti-seizure medicine works similarly well and more quickly when given through an IV or when given as a shot in the muscle. Two similar medicines will be used. Both are already used by paramedics in the field and by doctors in the hospital to stop seizures. One is commonly given by IV, and the other is commonly given as a shot in the muscle. In this study, the shot will be given using a device similar to an EpiPen-which is an autoinjector used by people with severe allergies.

Approximately 1,024 persons whose seizures are continuing after emergency medical service (EMS) arrival and who meet all eligibility criteria will be enrolled in the trial. Every participant will be treated with anti-seizure medicine by the paramedics. At random, half the participants will be in one group and half in another. Half the participants will receive the study medicine through an IV and will be given a shot in the muscle without medicine (placebo). The other half will receive the medicine as a shot in the muscle plus an IV without medicine (placebo).

In September 2010, more rapid than expected enrollment made it feasible to increase the sample size of the study from 800 to 1,024 with the already available funding. The goals of the expansion were to enroll more pediatric subjects (since the trial was enrolling slightly fewer than anticipated) and to improve the power of the study to 90%, which was initially desired. It is important to understand that the extended enrollment was not a sample size re-estimation in any way. The opportunity to extend the trial is pragmatic, based solely on the early enrollment success of the trial. It is not informed by the planned interim analyses that have been performed, the results of which remain sequestered, and there have been no unscheduled interim analyses. The firewall that prevents the blinded leadership from any knowledge of the outcome data has been diligently maintained throughout the process of proposing and implementing this extension.

ELIGIBILITY:
Inclusion Criteria:

* Paramedics or reliable witnesses verify 5 minutes of either continuous seizure activity or of repeated convulsive seizure activity where the patient does not regain consciousness (operationally defined as meaningful speech or obeying commands) between seizures.
* Patient is still seizing at the time of paramedic treatment with study medications.
* Estimated weight equal to or greater than 13 kg.
* Subject to be transported to a RAMPART participating hospital.

Exclusion Criteria:

* Major trauma as the precipitant of the seizure
* Hypoglycemia (as defined by local EMS protocol or a glucose < 60 mg/dL)
* Known allergy to midazolam or lorazepam
* Cardiac arrest or heart rate (HR) <40 beats per minute
* Sensitivity to benzodiazepines
* Medical alert tag marked with "RAMPART declined"
* Prior treatment of this seizure with diazepam autoinjector as part of another study
* Known pregnancy
* Prisoners

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1023 (Actual)
Dates: Start 2009-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Silbergleit, MD, Principal Investigator — University of Michigan; Daniel H Lowenstein, MD, Principal Investigator — University of California, San Francisco; Valerie L Durkalski, PhD, Principal Investigator — Medical University of South Carolina
Locations (17):
- United States (17):
  - University of Arizona, Tucson, Arizona
  - Stanford University, Palo Alto, California
  - University of California-San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - University of Kentucky, Lexington, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Wayne State University, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - New York Presbyterian Hospital, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania/York, Philadelphia, Pennsylvania
  - Temple University-Main Line, Philadelphia, Pennsylvania
  - University of Texas-Houston, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Sherman NA, Silbergleit R, Bengelink EM, Durkalski V, Wolter KD. The Midazolam RAMPART Study Medical Records Project: A Unique Use of Real-World Data in a Complex Collaborative Partnership to Support a New Drug Application. Ther Innov Regul Sci. 2023 Jan;57(1):132-141. doi: 10.1007/s43441-022-00447-4. Epub 2022 Aug 20. PMID 35987977
- [Derived] Silbergleit R, Lowenstein D, Durkalski V, Conwit R; NETT Investigators. Lessons from the RAMPART study--and which is the best route of administration of benzodiazepines in status epilepticus. Epilepsia. 2013 Sep;54 Suppl 6(0 6):74-7. doi: 10.1111/epi.12284. PMID 24001080
- [Derived] Silbergleit R, Biros MH, Harney D, Dickert N, Baren J; NETT Investigators. Implementation of the exception from informed consent regulations in a large multicenter emergency clinical trials network: the RAMPART experience. Acad Emerg Med. 2012 Apr;19(4):448-54. doi: 10.1111/j.1553-2712.2012.01328.x. PMID 22506949
- [Derived] Silbergleit R, Durkalski V, Lowenstein D, Conwit R, Pancioli A, Palesch Y, Barsan W; NETT Investigators. Intramuscular versus intravenous therapy for prehospital status epilepticus. N Engl J Med. 2012 Feb 16;366(7):591-600. doi: 10.1056/NEJMoa1107494. PMID 22335736
- [Derived] Silbergleit R, Lowenstein D, Durkalski V, Conwit R; Neurological Emergency Treatment Trials (NETT) Investigators. RAMPART (Rapid Anticonvulsant Medication Prior to Arrival Trial): a double-blind randomized clinical trial of the efficacy of intramuscular midazolam versus intravenous lorazepam in the prehospital treatment of status epilepticus by paramedics. Epilepsia. 2011 Oct;52 Suppl 8(Suppl 8):45-7. doi: 10.1111/j.1528-1167.2011.03235.x. PMID 21967361
- See also: RAMPART Study Public Information Web Site — http://rampart.umich.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects treated for status epilepticus in the prehospital setting by paramedics were enrolled at the scene between June 2009 and January 2011. A total of 1023 subject enrollments represented 893 unique subjects with a reenrollment rate of 13%. RAMPART involved 4314 paramedics, 33 EMS agencies, and 79 receiving hospitals across the United States.
Pre-assignment Details: Number of patients enrolled includes any repeat enrollments for those who presented to emergency medical services (EMS) with status epilepticus more than once. The number assigned to treatment in the intention-to-treat analysis includes every patient who was enrolled in the study but only the initial enrollment for those enrolled more than once.
Groups:
- Intramuscular (IM) Anticonvulsant: This group gets active treatment with an anticonvulsant by the intramuscular route of administration. IM administration by autoinjector of midazolam 5 mg for subjects under estimated weight of 40 kg or midazolam 10 mg for subjects with estimated weight of 40 kg or above, IV administration of matching volume of IV flush.
- Intravenous (IV) Anticonvulsant: This group gets active treatment with an anticonvulsant by the intravenous route of administration. IV administration of lorazepam 2 mg for subjects under estimated weight of 40 kg or midazolam 4 mg for subjects with estimated weight of 40 kg or above, IM administration by autoinjector of matching volume of saline.
Period: Overall Study
Arm/Group | Intramuscular (IM) Anticonvulsant | Intravenous (IV) Anticonvulsant
Started | 448 | 445
Completed | 448 | 445
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intramuscular (IM) Anticonvulsant | Intravenous (IV) Anticonvulsant | Total
Number analyzed (Participants) | 448 | 445 | 893
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (22) | 44 (22) | 43 (22)
Age, Customized [Number; unit: participants]
  0-5 years | 32 | 29 | 61
  6-10 years | 15 | 20 | 35
  11-20 years | 28 | 21 | 49
  21-40 years | 114 | 112 | 226
  41-60 years | 169 | 169 | 338
  >61 years | 90 | 94 | 184
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 198 | 207 | 405
  Male | 250 | 238 | 488
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 49 | 57 | 106
  Not Hispanic or Latino | 310 | 290 | 600
  Unknown or Not Reported | 89 | 98 | 187
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 5 | 8
  Asian | 8 | 14 | 22
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 229 | 224 | 453
  White | 165 | 183 | 348
  More than one race | 9 | 5 | 14
  Unknown or Not Reported | 32 | 13 | 45
Region of Enrollment [Number; unit: participants]
  United States | 448 | 445 | 893
Dose tier [Number; unit: participants] — All adults and those children with an estimated body weight of more than 40 kg received either 10 mg of intramuscular midazolam followed by intravenous placebo or intramuscular placebo followed by 4 mg of intravenous lorazepam. Children with an estimated weight of 13 to 40 kg received either 5 mg of intramuscular midazolam followed by intravenous placebo or intramuscular placebo followed by 2 mg of intravenous lorazepam.
  participants
    children with an estimated weight of 13 to 40 kg | 62 | 59 | 121
    Children estimated >40kg and All Adults | 386 | 386 | 772
History of epilepsy [Number; unit: participants]
  Yes | 293 | 295 | 588
  No | 111 | 103 | 214
  Not documented | 44 | 47 | 91
Final diagnosis [Number; unit: participants] — Determined by medical record review at the time of hospital discharge
  participants
    Status epilepticus | 404 | 399 | 803
    Nonepileptic spell | 31 | 32 | 63
    Undetermined | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Termination of Seizures at ED Arrival With no Rescue Therapy Given
Description: The primary outcome was termination of seizures before arrival in the emergency department (ED) without the need for the paramedics to provide rescue therapy. Subjects did not reach the primary outcome if they were having seizures on arrival in the emergency department or if they received rescue medication before arrival. Termination of seizures on arrival was determined according to the clinical judgment of the attending emergency physician and was based on examination of the subjects, their clinical course, and results of any routine diagnostic testing.
Time Frame: Duration of prehospital care, outcome is determined upon arrival at the ED on the day of enrollment (average 20 minutes).
Measure: Number; unit: participants
Groups:
- IM Midazolam: Subjects in whom the study IM autoinjector contained active treatment with midazolam
- IV Lorazepam: Subjects in whom the study IV infusion contained active treatment with lorazepam
Arm/Group | IM Midazolam | IV Lorazepam
Number analyzed (Participants) | 448 | 445
participants | 329 | 282
Statistical Analysis 1: Comparison: IM Midazolam vs IV Lorazepam; The null hypothesis of inferiority was tested with a one-sided z statistic. Sample size was estimated assuming independent proportions, 2 interim analyses, 70% control event rate; 90% power; a noninferiority margin of 10%; and a 1-sided test with type I error probability of 0.025. A sample size of 890 (445 per treatment group) was inflated by 15% (1024 subjects) to account for inadvertent repeated enrollment of the same subjects. Repeated enrollments of the same subject were not analyzed; Test type: Non-Inferiority or Equivalence — Assay sensitivity established by extensive review of lorazepam efficacy data. Noninferiority margin of 10% established by both clinical and statistical reasoning; p < 0.001, one-sided z statistic; Risk Difference (RD) = 0.10, 95% CI 2-sided [0.04 to 0.16]

2. Secondary Outcome: Number of Subjects With Endotracheal Intubation Within 30 Min After ED Arrival
Description: Endotracheal intubation performed or attempted by EMS or within 30 minutes after ED arrival is abstracted from the ED record physician and nursing records. Endotracheal intubation includes placement of a definitive tracheal airway (oro-, naso-, cricothyroidotomy, or tracheostomy) for support of respirations or protection of airway. Non-definitive and/or non-tracheal airways (oral or nasal airways, laryngeal mask airways, or esophageal obturator airways) are not included if the patient is not subsequently intubated unless specifically deemed to have been used in lieu of tracheal intubation.
Time Frame: anytime before 30 minutes after ED arrival
Measure: Number; unit: participants
Arm/Group | IM Midazolam | IV Lorazepam
Number analyzed (Participants) | 448 | 445
participants | 63 | 64
Statistical Analysis 1: Comparison: IM Midazolam vs IV Lorazepam; Test type: Superiority or Other; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.70 to 1.34]

3. Secondary Outcome: Number of Subjects Hospitalized
Description: Hospital and ICU admission from the ED, and length of stay, is abstracted from the hospital admission record. ICU admission is recorded as occurring only if the ICU is the initial inpatient unit for the patient.
Time Frame: at ED disposition on day of enrollment
Measure: Number; unit: participants
Arm/Group | IM Midazolam | IV Lorazepam
Number analyzed (Participants) | 448 | 445
participants | 258 | 292
Statistical Analysis 1: Comparison: IM Midazolam vs IV Lorazepam; Test type: Superiority or Other; Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.79 to 0.98]

4. Secondary Outcome: Number of Subjects Admitted to an Intensive Care Unit (ICU)
Description: as for outcome 3
Time Frame: at time of disposition on day of enrollment
Measure: Number; unit: participants
Arm/Group | IM Midazolam | IV Lorazepam
Number analyzed (Participants) | 448 | 445
participants | 128 | 161
Statistical Analysis 1: Comparison: IM Midazolam vs IV Lorazepam; Test type: Superiority or Other; Risk Ratio (RR) = 0.79, 95% CI 2-sided [0.65 to 0.95]

5. Secondary Outcome: Number of Subjects With Recurrent Seizure Within 12 Hours After ED Arrival
Description: Acute seizure recurrence is defined as any further convulsive or electrographic seizures occurring in the first 12 hours of hospitalization, if they require additional antiepileptic medications, in subjects that had been determined not to be having seizures on ED arrival.
Time Frame: within 12 hours after ED arrival
Measure: Number; unit: participants
Arm/Group | IM Midazolam | IV Lorazepam
Number analyzed (Participants) | 448 | 445
participants | 51 | 47
Statistical Analysis 1: Comparison: IM Midazolam vs IV Lorazepam; All participants were included in this analysis of rate of recurrence because this is the most clinically relevant denominator, although, by definition, only participants who stopped could have recurrent seizures; Test type: Superiority or Other; Risk Ratio (RR) = 1.08, 95% CI 2-sided [0.74 to 1.56]

6. Secondary Outcome: Number of Subjects With Hypotension
Description: Acute hypotension is defined as a systolic blood pressure of < 90 mmHg sustained for greater than 5 minutes and for which the patient was treated with a continuous IV infusion of a vasopressor.
Time Frame: participants were followed for the duration of hospital stay, an average of 6 days
Measure: Number; unit: participants
Arm/Group | IM Midazolam | IV Lorazepam
Number analyzed (Participants) | 448 | 445
participants | 12 | 13
Statistical Analysis 1: Comparison: IM Midazolam vs IV Lorazepam; Test type: Superiority or Other; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.42 to 1.98]

7. Secondary Outcome: Number of Subjects With IM Injection-site Complications
Description: IM injection site complications are defined as any symptoms or signs of injury or reaction at the site of the study IM injection requiring treatment. This includes extensive hematoma requiring treatment (decompression, pressure dressings, or discontinuation of anticoagulant or antithrombotic medications). Treatment does not include imaging without other interventions. This definition also includes wound infection requiring antibiotic therapy, retained foreign bodies requiring exploration and removal, or other similar wound problems.
Time Frame: participants were followed for the duration of hospital stay, an average of 6 days
Measure: Number; unit: participants
Arm/Group | IM Midazolam | IV Lorazepam
Number analyzed (Participants) | 448 | 445
participants | 4 | 2
Statistical Analysis 1: Comparison: IM Midazolam vs IV Lorazepam; Test type: Superiority or Other; Risk Ratio (RR) = 1.99, 95% CI 2-sided [0.30 to 10.70]

8. Secondary Outcome: Number of Subjects With IV Injection-site Complications
Description: IV insertion site complications are defined as any symptoms or signs of injury or reaction at the site of the study IV placed by paramedics and used for study medication. This includes thrombosis, phlebitis, or skin infection requiring specific treatment including compresses, antibiotics, or wound care.
Time Frame: participants were followed for the duration of hospital stay, an average of 6 days
Measure: Number; unit: participants
Arm/Group | IM Midazolam | IV Lorazepam
Number analyzed (Participants) | 448 | 445
participants | 0 | 3

9. Secondary Outcome: Length of Intensive Care Unit (ICU) Stay in Days
Description: Continuous days of initial ICU stay from time of admission
Time Frame: participants were followed for the duration of hospital stay, an average of 6 days
Population: All participants with ICU length of stay data
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IM Midazolam | IV Lorazepam
Number analyzed (Participants) | 123 | 155
days | 5.7 (9.5) | 4.1 (4.7)
Statistical Analysis 1: Comparison: IM Midazolam vs IV Lorazepam; Test type: Superiority or Other; p = 0.09, t-test, 2 sided

10. Secondary Outcome: Length of Hospital Stay in Days
Description: Continuous acute care inpatient hospital days from day of admission until discharge
Time Frame: participants were followed for the duration of hospital stay, an average of 6 days
Population: All subjects with hospital length of stay data
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IM Midazolam | IV Lorazepam
Number analyzed (Participants) | 251 | 285
days | 6.7 (10.0) | 5.5 (6.4)
Statistical Analysis 1: Comparison: IM Midazolam vs IV Lorazepam; Test type: Superiority or Other; p = 0.11, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected through subject end of study (emergency department or hospital discharge).
Description: Number of participants at risk includes every enrollment (including repeat enrollments in some subjects). This reflects the number of interventions given.
Arm/Group | IM Midazolam | IV Lorazepam
Serious Adverse Events (participants affected / at risk) | 137/514 | 156/509
Other Adverse Events (participants affected / at risk) | 103/514 | 95/509
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IM Midazolam (N=514) | IV Lorazepam (N=509)
Depressed level of consciousness (Nervous system disorders) | 49 | 45
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 33 | 51
Convulsion (Nervous system disorders) | 33 | 39
Mental status changes (Nervous system disorders) | 9 | 10
Sepsis/SIRS/organ failure (Infections and infestations) | 8 | 8
Pneumonia/ Aspiration pneumonia (Infections and infestations) | 2 | 11
Myocardial infarction (Cardiac disorders) | 5 | 7
Hypotension (Cardiac disorders) | 5 | 7
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 5 | 5
Alcohol/Drug withdrawal syndrome (General disorders) | 5 | 5
Cerebral hemorrhage (Nervous system disorders) | 4 | 0
Renal failure, acute (Renal and urinary disorders) | 4 | 0
Ischemic stroke (Nervous system disorders) | 2 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 3
Hypoglycemia (Endocrine disorders) | 2 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Hypothermia (General disorders) | 0 | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 2
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Brain mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 1
Pulmonary embolism (Vascular disorders) | 1 | 1
Chest pain (General disorders) | 1 | 0
Delirium (Nervous system disorders) | 1 | 0
Hematoma (General disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Hyperglycemic hyperosmolar nonketotic syndrome (Endocrine disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Subarachnoid hemorrhage (Nervous system disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Transfusion reaction (Blood and lymphatic system disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Pseudoseizures (Psychiatric disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypertension (Cardiac disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Post-extubation stridor/airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Psychosis (Psychiatric disorders) | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 1
Vomiting/Nausea (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IM Midazolam (N=514) | IV Lorazepam (N=509)
Convulsion (Nervous system disorders) | 45 | 38
Mental status changes (Nervous system disorders) | 20 | 20
Vomiting/Nausea (Gastrointestinal disorders) | 15 | 23
Pyrexia (General disorders) | 23 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No